CLINICAL TRIAL: NCT02981680
Title: Effect of Remote Ischemic Preconditioning on the Incidence of Acute Kidney Injury in Patients Undergoing Coronary Artery Bypass Graft Surgery: A Randomized Controlled Trial
Brief Title: Effect of Remote Ischemic Preconditioning on the Incidence of Acute Kidney Injury in Patients Undergoing Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sina Bagheri, Principal Investigator, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 94-01-01-11214
Record Dates: First submitted 2016-11-28; First posted 2016-12-05 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Acute Kidney Injury; Coronary Artery Bypass; Ischemic Preconditioning
Keywords: remote ischemic preconditioning; transient limb ischemia; acute kidney injury; coronary artery bypass graft surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- RIPC (Experimental): Patients in the remote ischemic preconditioning (RIPC) group will receive three sequential sphygmomanometer cuff inflations on their right upper arm after induction of anesthesia in the operating room. The cuff will be inflated by the OR nurse up to 200 mmHg for five minutes each occasion, with five minutes deflation in between inflations. Following this pre-conditioning phase, surgery will be started. The entire pre-conditioning phase will last 30 minutes.
  Interventions: Procedure: Remote Ischemic Preconditioning (RIPC)
- sham-RIPC (Sham Comparator): Patients in the sham-RIPC group will have the sphygmomanometer cuff placed on their right upper arm, but the cuff will not be inflated. Similar to patients in the RIPC group, patients in the sham-RIPC group will undergo the same 30 minute delay before starting surgery.
  Interventions: Procedure: sham-RIPC

INTERVENTIONS:
Procedure: Remote Ischemic Preconditioning (RIPC) — Remote ischemic preconditioning (RIPC) is a phenomenon in which brief ischemia of one organ or tissue, provokes a protective effect that can reduce the mass of infarction caused by vessel occlusion and reperfusion.
  Arms: RIPC
Procedure: sham-RIPC
  Arms: sham-RIPC

SUMMARY:
Background:

Acute kidney injury (AKI) following coronary artery bypass graft (CABG) surgery is a major complication occurring in 1% to 53% of patients (depending on how it is defined) with the pooled rate of 18.2% and unfortunately 2.1% of them require renal replacement therapy. Cardiopulmonary bypass (CPB)-associated AKI increases mortality 2-4 fold regardless of AKI definition. It is also associated with increased risk of postoperative stroke, acute myocardial infarction, cardiac tamponade, heart failure, and lengthened intensive care unit and hospital stays. Even minor elevations of postoperative serum creatinine (SCr) have been associated with a significant increase in 30-day mortality, from a 3-fold increase risk for a small elevation of up to 0.5 mg/dL from baseline to an 18-fold increase risk of death with a SCr rise greater than 0.5 mg/dL.

The pathogenesis of CPB-associated AKI is complicated and includes hemodynamic, inflammatory and other mechanisms that interact at a cellular level. To date, despite several clinical trials of pharmacologic interventions, none of them have demonstrated conclusively efficacy in the prevention of AKI after cardiac surgery.

Remote ischemic preconditioning (RIPC) is a phenomenon in which brief ischemia of one organ or tissue, provokes a protective effect that can reduce the mass of infarction caused by vessel occlusion and reperfusion. In CABG surgery, cardiomyocyte injury caused by myocardial protection failure is predominantly responsible for adverse outcomes. RIPC was shown to reduce troponin release 24 h postoperatively in children undergoing corrective surgery for congenital heart disease. Other studies demonstrated that RIPC using brief ischemia and reperfusion of the upper limb reduces myocardial injury in adult patients undergoing CABG surgery.

Due to the similarities between the mechanisms of ischemia-reperfusion injury produced by RIPC and those proposed for AKI after CPB, we decided to test the hypothesis that RIPC prevents AKI in patients undergoing CABG surgery.

Methods:

180 patients who fulfill all inclusion and exclusion criteria will be divided into case and control groups (90 patients in the case and 90 patients in the control group).

Patients in the treatment group will receive three sequential sphygmomanometer cuff inflations on their right upper arm after induction of anesthesia in the operating room. The cuff will be inflated by the OR nurse up to 200 mmHg for five minutes each occasion, with five minutes deflation in between inflations. Following this pre-conditioning phase, surgery will be started. The entire pre-conditioning phase will last 30 minutes.

Patients in the control group will have the sphygmomanometer cuff placed on their right upper arm, but the cuff will not be inflated. Similar to patients in the treatment group, patients in the control group will undergo the same 30 minute delay before starting surgery.

Complete blood count (CBC), SCr, liver function test (LFT), will be checked before surgery.

After surgery, SCr will be checked daily. If AKI occurs, it will be managed and dialysis will be done if the patient requires it. All patients will undergo electrocardiogram and LFT after CABG surgery during hospital course.

ELIGIBILITY:
Inclusion Criteria:

* Candidate cardiac surgical patients
* Elective or urgent on pump coronary artery bypass grafting (CABG)
* Age 18 to 85 years
* Signed informed consent

Exclusion Criteria:

* End-stage renal disease (receiving hemodialysis or glomerular filtration rate <15 ml/min/1.73m2)
* Peripheral vascular disease
* Severe hepatic disease
* Planned off-pump surgery
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative acute kidney injury (AKI) | Within the first 72 hours after surgery
  Defined as an elevation of serum creatinine of ≥0.3 mg/dl or ≥50% within 72 hours after surgery

SECONDARY OUTCOMES:
Duration of hospital stay | Through hospital stay after surgery, an average of 5 days
Duration of ICU stay | Through ICU stay, an average of 3 days
All cause mortality | Through hospital stay after surgery, an average of 5 days
Number of participants requiring dialysis | Through hospital stay after surgery, an average of 5 days
Postoperative liver function | Preoperatively and at 24 h post-surgery
  By measuring serum aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin (TBIL), and albumin
Incidence of postoperative atrial fibrillation (AF) | Within the first 72 hours after surgery
  Defined as the incidence of new-onset AF lasting for five minutes or longer
Incidence of postoperative stroke | Through hospital stay after surgery, an average of 5 days
  Defined as a new ischemic or hemorrhagic cerebrovascular accident with neurological deficit lasting >24 h

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Mahdi Sagheb, MD, Study Chair — Department of Nephrology, Shiraz University of Medical Sciences, Shiraz, Iran
Locations (1):
- Shiraz University of Medical Sciences, Shiraz, Fars, Iran

REFERENCES:
- [Background] Pickering JW, James MT, Palmer SC. Acute kidney injury and prognosis after cardiopulmonary bypass: a meta-analysis of cohort studies. Am J Kidney Dis. 2015 Feb;65(2):283-93. doi: 10.1053/j.ajkd.2014.09.008. Epub 2014 Nov 5. PMID 25445101
- [Background] Karkouti K, Wijeysundera DN, Yau TM, Callum JL, Cheng DC, Crowther M, Dupuis JY, Fremes SE, Kent B, Laflamme C, Lamy A, Legare JF, Mazer CD, McCluskey SA, Rubens FD, Sawchuk C, Beattie WS. Acute kidney injury after cardiac surgery: focus on modifiable risk factors. Circulation. 2009 Feb 3;119(4):495-502. doi: 10.1161/CIRCULATIONAHA.108.786913. Epub 2009 Jan 19. PMID 19153273
- [Background] Gallagher S, Jones DA, Lovell MJ, Hassan S, Wragg A, Kapur A, Uppal R, Yaqoob MM. The impact of acute kidney injury on midterm outcomes after coronary artery bypass graft surgery: a matched propensity score analysis. J Thorac Cardiovasc Surg. 2014 Mar;147(3):989-95. doi: 10.1016/j.jtcvs.2013.03.016. Epub 2013 Apr 12. PMID 23587469
- [Background] Ryden L, Ahnve S, Bell M, Hammar N, Ivert T, Holzmann MJ. Acute kidney injury following coronary artery bypass grafting: early mortality and postoperative complications. Scand Cardiovasc J. 2012 Apr;46(2):114-20. doi: 10.3109/14017431.2012.657229. Epub 2012 Feb 10. PMID 22324648
- [Background] Mehta RH, Honeycutt E, Patel UD, Lopes RD, Shaw LK, Glower DD, Harrington RA, Califf RM, Sketch MH Jr. Impact of recovery of renal function on long-term mortality after coronary artery bypass grafting. Am J Cardiol. 2010 Dec 15;106(12):1728-34. doi: 10.1016/j.amjcard.2010.07.045. Epub 2010 Oct 26. PMID 21126617
- [Background] Loef BG, Epema AH, Smilde TD, Henning RH, Ebels T, Navis G, Stegeman CA. Immediate postoperative renal function deterioration in cardiac surgical patients predicts in-hospital mortality and long-term survival. J Am Soc Nephrol. 2005 Jan;16(1):195-200. doi: 10.1681/ASN.2003100875. Epub 2004 Nov 24. PMID 15563558
- [Background] Olsson D, Sartipy U, Braunschweig F, Holzmann MJ. Acute kidney injury following coronary artery bypass surgery and long-term risk of heart failure. Circ Heart Fail. 2013 Jan;6(1):83-90. doi: 10.1161/CIRCHEARTFAILURE.112.971705. Epub 2012 Dec 10. PMID 23230310
- [Background] Dasta JF, Kane-Gill SL, Durtschi AJ, Pathak DS, Kellum JA. Costs and outcomes of acute kidney injury (AKI) following cardiac surgery. Nephrol Dial Transplant. 2008 Jun;23(6):1970-4. doi: 10.1093/ndt/gfm908. Epub 2008 Jan 4. PMID 18178605
- [Background] Lassnigg A, Schmidlin D, Mouhieddine M, Bachmann LM, Druml W, Bauer P, Hiesmayr M. Minimal changes of serum creatinine predict prognosis in patients after cardiothoracic surgery: a prospective cohort study. J Am Soc Nephrol. 2004 Jun;15(6):1597-605. doi: 10.1097/01.asn.0000130340.93930.dd. PMID 15153571
- [Background] Rosner MH, Okusa MD. Acute kidney injury associated with cardiac surgery. Clin J Am Soc Nephrol. 2006 Jan;1(1):19-32. doi: 10.2215/CJN.00240605. Epub 2005 Oct 19. PMID 17699187
- [Background] Burns KE, Chu MW, Novick RJ, Fox SA, Gallo K, Martin CM, Stitt LW, Heidenheim AP, Myers ML, Moist L. Perioperative N-acetylcysteine to prevent renal dysfunction in high-risk patients undergoing cabg surgery: a randomized controlled trial. JAMA. 2005 Jul 20;294(3):342-50. doi: 10.1001/jama.294.3.342. PMID 16030279
- [Background] Young EW, Diab A, Kirsh MM. Intravenous diltiazem and acute renal failure after cardiac operations. Ann Thorac Surg. 1998 May;65(5):1316-9. doi: 10.1016/s0003-4975(98)00157-x. PMID 9594859
- [Background] Ranucci M, Soro G, Barzaghi N, Locatelli A, Giordano G, Vavassori A, Manzato A, Melchiorri C, Bove T, Juliano G, Uslenghi MF. Fenoldopam prophylaxis of postoperative acute renal failure in high-risk cardiac surgery patients. Ann Thorac Surg. 2004 Oct;78(4):1332-7; discussion 1337-8. doi: 10.1016/j.athoracsur.2004.02.065. PMID 15464494
- [Background] Venugopal V, Ludman A, Yellon DM, Hausenloy DJ. 'Conditioning' the heart during surgery. Eur J Cardiothorac Surg. 2009 Jun;35(6):977-87. doi: 10.1016/j.ejcts.2009.02.014. Epub 2009 Mar 25. PMID 19324569
- [Background] Cheung MM, Kharbanda RK, Konstantinov IE, Shimizu M, Frndova H, Li J, Holtby HM, Cox PN, Smallhorn JF, Van Arsdell GS, Redington AN. Randomized controlled trial of the effects of remote ischemic preconditioning on children undergoing cardiac surgery: first clinical application in humans. J Am Coll Cardiol. 2006 Jun 6;47(11):2277-82. doi: 10.1016/j.jacc.2006.01.066. Epub 2006 May 15. PMID 16750696
- [Background] Hausenloy DJ, Mwamure PK, Venugopal V, Harris J, Barnard M, Grundy E, Ashley E, Vichare S, Di Salvo C, Kolvekar S, Hayward M, Keogh B, MacAllister RJ, Yellon DM. Effect of remote ischaemic preconditioning on myocardial injury in patients undergoing coronary artery bypass graft surgery: a randomised controlled trial. Lancet. 2007 Aug 18;370(9587):575-9. doi: 10.1016/S0140-6736(07)61296-3. PMID 17707752
- [Background] Venugopal V, Hausenloy DJ, Ludman A, Di Salvo C, Kolvekar S, Yap J, Lawrence D, Bognolo J, Yellon DM. Remote ischaemic preconditioning reduces myocardial injury in patients undergoing cardiac surgery with cold-blood cardioplegia: a randomised controlled trial. Heart. 2009 Oct;95(19):1567-71. doi: 10.1136/hrt.2008.155770. Epub 2009 Jun 8. PMID 19508973
- [Background] Bonventre JV, Zuk A. Ischemic acute renal failure: an inflammatory disease? Kidney Int. 2004 Aug;66(2):480-5. doi: 10.1111/j.1523-1755.2004.761_2.x. PMID 15253693
- [Background] Yellon DM, Hausenloy DJ. Myocardial reperfusion injury. N Engl J Med. 2007 Sep 13;357(11):1121-35. doi: 10.1056/NEJMra071667. No abstract available. PMID 17855673